CLINICAL TRIAL: NCT06242912
Title: Evidence Development in Cancer Treatment - Real World: PREDiCTrw
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: British Columbia Cancer Agency (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: PREDiCTrw
Record Dates: First submitted 2024-01-22; First posted 2024-02-05 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Therapy (Experimental): Regular disease assessment (eg radiographic imaging) and quality of life (QOL) questionnaires
  Interventions: Behavioral: QOL - quality of life; Diagnostic Test: Radiographic or laboratory evaluation

INTERVENTIONS:
Behavioral: QOL - quality of life — QOL assessments using EQ5D (Euroqol 5 dimension) +/- ESAS (Edmonton Symptom Assessment Scale) +/- CPC (Canadian Problem Checklist) every 4-8 weeks +/- 2 weeks
Diagnostic Test: Radiographic or laboratory evaluation — Radiographic or laboratory evaluation every 12 weeks +/- 2 weeks

SUMMARY:
This pilot clinical trial aims to assess the real world quality of life and survival of patients treated with therapy that has preliminary evidence of efficacy but uncertainty of the magnitude of clinical benefit or cost effectiveness in subjects with cancer. The goal of this study is to collect real world evidence with respect to quality of life and outcomes to support decision making.

DETAILED DESCRIPTION:
Clinical practice involves incorporating new data into treatment recommendations including non randomized phase I/II studies. Clinicians' decision-making is swayed by alternative endpoints like response rate (RR), depth of response and progression free survival (PFS), presumed to be surrogates for overall survival (OS). Determination of the added value of these new therapies in terms of outcomes and quality of life (QOL) is challenging in the absence of comparators in trials resulting in increased uncertainty in terms of outcomes, quality of life and cost-effectiveness.

With the possibility of a randomized clinical trial evidence being low in certain populations, the use of real world data (RWD) can provide information regarding therapies with preliminary evidence of efficacy but uncertainty of the magnitude of clinical benefit or cost effectiveness. With RWD, patients may receive access to therapies and participate in the evidence generation package.

This study proposes to use RWD to generate evidence to evaluate therapies with preliminary evidence of efficacy but uncertainty of the magnitude of clinical benefit or cost effectiveness. The key components include regular interval disease assessments (eg radiographic imaging) and collection of patient reported outcomes (PROs) using standardized QOL questionnaires. The aim is to provide high quality real world evidence (RWE) for assessment and economic modelling to reduce uncertainty and facilitate decision-making.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with cancer for which there remains ongoing questions regarding clinical effectiveness and/or cost effectiveness regarding a therapeutic agent
* Eastern Co-operative Group (ECOG) 0-2
* Life expectancy of at least 12 weeks
* Adequate hematologic and end organ function for drug treatment per the clinician's assessment
* Asymptomatic or treated brain metastases permitted
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods that result in a failure rate of less than 1% per year during the treatment period and for at least 5 months after the last dose.
* For men: agreement to remain abstinent (refrain from heterosexual intercourse with a female partner of childbearing potential or who is pregnant) or use contraceptive measures, and agreement to refrain from donating sperm, during the treatment period and for at least 5 months after the last dose.
* Ability to give informed consent for the study procedures defined in this protocol.

Exclusion Criteria:

* Treatment with any approved or investigational agent or participation in another clinical trial with therapeutic intent within 14 days prior to enrollment.
* Inability to complete quality of life questionnaires
* Pregnancy or breastfeeding.
* Any significant cardiovascular disease, comorbidity (i.e. recent major infection, HIV, tuberculosis) or major surgical procedure within 21 days that in the opinion of the investigator renders the proposed treatment unsafe.
* Subjects who are otherwise felt by the treating clinician to be unfit to proceed with this protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-01-22 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival | From date of initiation until the date of death from any cause, whichever came first, assessed up to 100 months
  Overall survival from initiation of therapy

SECONDARY OUTCOMES:
Response rate | From date of initiation until the date of death from any cause, whichever came first, assessed up to 100 months
  Response rate as defined by standard measurement for tumor site (eg RECIST 1.1)
Progression/event free survival | From date of initiation until the date of progression or date of death from any cause, whichever came first, assessed up to 100 months
  Progression or event free survival from initiation of therapy
Quality of life assessments | From date of initiation until the date of death from any cause, whichever came first, assessed up to 100 months
  Quality of life assessments using EQ5D scale 1 to 5 with 5 being extreme problems
Quality adjust survival | From date of initiation until the date of death from any cause, whichever came first, assessed up to 100 months
  Quality adjusted survival from initiation of therapy
Physician assessed response rate | From date of initiation until the date of death from any cause, whichever came first, assessed up to 100 months
  Response rate as defined by physician assessed response

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl Ho, MD, Study Chair — BC Cancer
Locations (1):
- BC Cancer, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No